CLINICAL TRIAL: NCT02005237
Title: Randomized Controlled Trial Investigating the Effects of a Standardized Aerobic Exercise Intervention on Cognitive Function and Brain Connectivity in Relapsing-remitting Multiple Sclerosis
Brief Title: Exercise in Multiple Sclerosis: Effects on Cognitive Function and Brain Connectivity
Acronym: AERCONN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AERCONN; 031A130 (Other Grant/Funding Number: BMBF)
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Multiple Sclerosis
Keywords: Exercise; Cognition; Neuroimaging; Rehabilitation; Connectivity
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobic Exercise (12 Weeks) (Experimental): Aerobic exercise on a bicycle ergometer, tailored to the individual's level of fitness. Duration: 12 weeks with 2-3 sessions per week.
  Interventions: Behavioral: Aerobic Exercise
- Waitlist Control Group (No Intervention): No intervention (patients randomized to this group will be offered access to the training program after completion of the trial)

INTERVENTIONS:
Behavioral: Aerobic Exercise — 3-months exercise program tailored to the individual level of aerobic fitness. Patients will exercise on a bicycle ergometer (2-3 session per week) according to a predefined training plan with increasing duration and intensity
  Arms: Aerobic Exercise (12 Weeks)

SUMMARY:
Cognitive dysfunction is frequent in patients with multiple sclerosis (MS) and to date, there are no available treatments to improve cognition in this patient population. Some evidence from animal studies and small clinical trials suggest that aerobic exercise might beneficially affect cognitive function in MS. The aim of this randomized-controlled trial is to explore if an aerobic exercise training program can enhance cognition in MS. In addition, we will employ neuroimaging markers to determine if exercise alters measures of brain structure and function.

Patients will be randomly assigned to either a 3-months exercise program (bicycle ergometry, 2-3 session per week) or a waitlist control group. The primary endpoint of the study is a test of verbal learning and memory. Secondary endpoints include neuroimaging markers of functional and structural connectivity in the brain. We hypothesize that exercise will improve verbal learning and memory and beneficially affect measures of brain connectivity.

DETAILED DESCRIPTION:
Background: Cognitive dysfunction is frequent in patients with multiple sclerosis (MS) and to date, there are no available treatments to improve cognition in this patient population. Some evidence from animal studies and small clinical trials suggest that aerobic exercise might beneficially affect cognitive function in MS.

Aims: This study aims to explore the potential of an aerobic exercise program on brain structure and function in MS in a single-blind, randomized controlled phase IIa trial. We hypothesize that exercise will improve verbal learning and memory (primary endpoint) as well as induce changes in neuroimaging markers of structural and functional central nervous system (CNS) connectivity (secondary endpoints). Tertiary outcomes will include walking ability, motor function and coordination, as well as patient-based outcomes (depression, fatigue, and health-related quality of life).

Design: This is a single-blind, randomized, controlled phase IIa trial with a parallel group design comparing 3 months of standardized aerobic exercise training (bicycle ergometry) to a waitlist control group (superiority framework). The allocation ratio of exercise to waitlist control is 1:1 with a sample size of n=60.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-remitting multiple sclerosis according to McDonald criteria
* Currently in remission
* Disease duration < 10 years
* Low to moderate physical disability (EDSS 0-3.5)
* On stable immunotherapy (>3 months) or without any planned treatment for the next year

Exclusion Criteria:

* Patients who are not able to understand the study concept due to severe cognitive deficits or psychiatric comorbidity
* Patients currently taking psychoactive drugs
* Patients unable to undergo aerobic exercise training for medical reasons
* Patients with active disease or uncertain stability under current immunomodulatory therapy (as judged by the treating neurologist)
* Patients with implants or body modifications (e.g. dental implants, piercings, tattoos, pacemakers etc.) which might interfere with MEG and MRI assessments
* Patients unable to travel to the study center 2-3 times a week for the duration of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-12; Primary Completion 2016-05 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in Verbal Learning and Memory | Baseline and at Month 3 (end of intervention)
  Verbal Learning and Memory will be assessed with the Verbal Learning and Memory Test (VLMT)

SECONDARY OUTCOMES:
Change in Functional Connectivity | Baseline and at Month 3 (end of intervention)
  Functional connectivity of CNS networks will be assessed by resting-state functional magnetic resonance imaging (rs fMRI) and resting-state magnetoencephalography (rs MEG)
Change in Structural Connectivity | Baseline and at Month 3 (end of intervention)
  Structural connectivity and integrity of CNS networks will be assessed by diffusion tensor imaging (DTI) as well as measures of gray matter density using magnetic resonance imaging (MRI)
Change in Neuropsychological Function | Baseline and at Month 3 (end of intervention)
  Neuropsychological function will be assessed using a standardized battery covering the following domains: visuospatial learning and memory, attention, processing speed, working memory, and social cognition

OTHER OUTCOMES:
Change in Patient-Reported Outcomes | Baseline and at Month 3 (end of intervention)
  Patient-reported outcomes will be assessed for depressive symptoms (IDS-30SR), fatigue (FSMC), quality of life (HAQUAMS), and walking (MSWS-12)
Change in Walking Ability | Baseline and at Month 3 (end of intervention)
  Walking ability will be assessed using the six-minute-walk test (6MWT) as well as Actibelt accelerometry

CONTACTS AND LOCATIONS:
Overall Officials: Stefan M Gold, PhD, Principal Investigator — Center for Molecular Neurobiology, University Hospital Hamburg Eppendorf; Andreas K Engel, MD, Principal Investigator — Dept Neurophysiology, University Hospital Hamburg Eppendorf; Christoph Heesen, MD, Principal Investigator — Dept Neurology, University Hospital Hamburg Eppendorf; Guido Nolte, PhD, Principal Investigator — Dept Neurophysiology, University Hospital Hamburg Eppendorf; Karl-Heinz Schulz, MD, PhD, Principal Investigator — Dept Sports Medicine, University Hospital Hamburg Eppendorf
Locations (1):
- University Hospital Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Derived] Baquet L, Hasselmann H, Patra S, Stellmann JP, Vettorazzi E, Engel AK, Rosenkranz SC, Poettgen J, Gold SM, Schulz KH, Heesen C. Short-term interval aerobic exercise training does not improve memory functioning in relapsing-remitting multiple sclerosis-a randomized controlled trial. PeerJ. 2018 Dec 12;6:e6037. doi: 10.7717/peerj.6037. eCollection 2018. PMID 30581662